CLINICAL TRIAL: NCT04021966
Title: Use of Fractional CO2 Laser for the Treatment of Vulvovaginal Atrophy: a Double-blinded Randomized Placebo-controlled Clinical Trial.
Acronym: CO2VVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: prof. dr. Jan Deprest (Other)
Responsible Party: Sponsor-Investigator, prof. dr. Jan Deprest, Professor, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S61680
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): In this arm, participants will have 3 real laser treatments first, followed by 3 consecutive sham treatments.
  Interventions: Procedure: Vaginal laser application
- Sham (Sham Comparator): In this arm, participants will have 3 sham treatments first, followed by 3 consecutive real laser treatments.
  Interventions: Procedure: Vaginal laser application

INTERVENTIONS:
Procedure: Vaginal laser application — One laser treatment cycle consists of 3 vaginal laser applications with a 4-weeks interval. Each application lasts around 5 minutes.
  The vaginal laser procedure will be performed in an outpatient setting, not requiring any specific preparation, analgesia or anesthesia, by one of two experienced operators.
  A vaginal probe will be gently inserted and manually rotated to provide a 360° treatment of the vaginal mucosa.

SUMMARY:
Purpose of the trial is to study the efficacy of fractional laser in alleviating genitourinary symptoms in menopausal women.

Primary outcome of the study is the efficacy of the laser procedure, intended as the amelioration of the severity of most bothersome symptom (MBS).

Therefore we conducted a single center, double-blinded randomized placebo-controlled cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

Healthy women with menopausal status (>1 year amenorrhea) AND with moderate to severe symptoms of VVA as measured by the MBS score ≥2.

Exclusion Criteria:

* Acute or recurrent urogenital infections
* Prolapse ≥ grade 3 according to the Pelvic Organ Prolapse Quantification System
* Hormonal replacement therapy within the last 6 months before study entry
* Use of local estrogens, moisturizers, lubricants or homeopathic preparations within the last 3 months
* Pelvic floor physiotherapy for pelvic floor disorders within the last 3 months
* Any condition that could interfere with study compliance

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure is the change in severity of most bothersome symptom (MBS) | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  The MBS is derived from a selected list of symptoms (consisting of the four most common symptoms of vaginal dryness, vaginal itching/irritation, vaginal soreness and dyspareunia). At baseline, participants are instructed to rate each of these symptoms as not present, mild, moderate or severe and then are asked to select a single symptom among those classified as moderate or severe as the MBS. The MBS is then followed through to the end of treatment, and the change in its severity is used to evaluate symptomatic improvement.

SECONDARY OUTCOMES:
Assessment of the effect of treatment on the female urogenital health, by means of the globally validated "Vaginal Health Index Score" (VHIS). | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  The VHIS includes scoring of vaginal moisture, vaginal fluid volume, vaginal elasticity, vaginal pH, and vaginal epithelial integrity on a scale of 1 (poorest) to 5 (best) according to the methods of Robert Wood Johnson Medical School. The lower the score, the greater the atrophy.
Assessment of the effect of treatment on the female urogenital health, by means of vaginal pH measurements. | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  Measurement of the vaginal pH is considered useful, effective, and inexpensive19. Studies have shown that a vaginal pH greater than 5.0 is associated with decreased serum estradiol and menopause. The vaginal pH will be measured with the use of a pH indicator strip and should be sampled from the lateral vaginal wall. This technique is validated. Such strips are available in every clinic.
Assessment of the effect of treatment on VVA symptoms (vaginal dryness, vaginal burning, vaginal itching, dyspareunia and dysuria) using the Visual Analog Scale (0-10cm, continuous scale). | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  For this measurement a continuous Visual Analogue Scale (0-10cm) is used (0 is no pain, 10 is the maximum pain score).
Assessment of the rate of patient satisfaction by means of the Patient Global Impression of Improvement (PGI), using a 5-point Likert scale (1=much worse, 2=worse, 3=same, 4=better, 5=much better). | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
Assessment of the degree of discomfort of the treatment procedure by the patient, by mean of a VAS-score(0-10cm, continuous scale). | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  For this measurement a continuous Visual Analogue Scale (0-10cm) is used (0 is no pain, 10 is the maximum pain score).
Assessment of the degree of difficulty encountered by the physician in performing the treatment, by means of a 5-point Likert scale (1=very difficult, 2=difficult, 3=neutral, 4=easy, 5=very easy). | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
Assessment of the long term satisfaction with, and the longevity of the effect of laser therapy, measured by the need for, and the timing for repeating the same, or initiating an alternative therapy. | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
Assessment of the vaginal wall thickness using in vivo microscopy (vaginal focal depth measurement). | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  VVA is associated with thinning of the vaginal epithelial layer due to the declining levels of circulating estrogen associated with VVA. Therefore, measurement of the vaginal wall thickness offers an objective measure in the diagnosis and evaluation of VVA and its treatment24. Vaginal focal depth measurements will be performed using the Cytocam-Incident Dark Field device (IDF), a validated technique to quantitatively assess vaginal microcirculation25. As part of the pelvic examination, the handheld device, covered with a sterile disposable cap, will gently be placed into contact with the anterior vaginal wall, 3cm above the hymen, assessing the distance between the subepithelial microcirculation and the epithelial surface in micrometers.
  At all clinical visits baseline/study parameters will be assessed before treatment and procedure related outcomes will be assessed after the procedure.
Effect of treatment, in sexually active patients, on female sexual function, by means of the validated "Female Sexual Function Index" (FSFI) specific questionnaire | Will be measured at baseline and during every next visit (vaginal applications and follow-up visits); ie. 0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 3 months, 6 months and 12 months post treatment
  The FSFI is a brief, 19-item self-report measure of female sexual function that provides scores on six domains of sexual function as well as a total score. The six domains include: desire (2 items; score range 1-5; factor 0.6; minimum score 1.2; maximum score 6.0), arousal (4 items; score range 0-5; factor 0.3; minimum score 0; maximum score 6.0), lubrication (4 items; score range 0-5; factor 0.3; minimum score 0; maximum score 6.0), orgasm (3 items; score range 0-5; factor 0.4; minimum score 0; maximum score 6.0), satisfaction (3 items; score range 0-5; factor 0.4; minimum score 0; maximum score 6.0), and pain (3 items; score range 0-5; factor 0.4; minimum score 0; maximum score 6.0).
  Full Scale Score Range: minimum score 2.0, maximum score 36.0. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page AS, Verbakel JY, Verhaeghe J, Latul YP, Housmans S, Deprest J. Laser versus sham for genitourinary syndrome of menopause: A randomised controlled trial. BJOG. 2023 Feb;130(3):312-319. doi: 10.1111/1471-0528.17335. Epub 2022 Nov 15. PMID 36349391